CLINICAL TRIAL: NCT00702702
Title: A Multi-Center, Placebo Controlled, Safety and Efficacy Study of the Selective Progesterone Receptor Modulator Proellex® (CDB-4124) in Anemic, Pre-Menopausal Women With Symptomatic Uterine Fibroids Requiring Hysterectomy
Brief Title: Safety and Efficacy of Proellex in Pre-menopausal Anemic Women With Symptomatic Uterine Fibroids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Repros stopped study for safety and FDA put study on hold because of safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZPU-301
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids; Anemia
Keywords: Uterine fibroids; Anemia
MeSH Terms: conditions — Leiomyoma; Anemia | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A 25 mg (Experimental): Proellex 25 mg, 1 - 25 mg capsule and 1 placebo capsule daily for 3 months
  Interventions: Drug: Proellex 25 mg
- B 50 mg (Experimental): Proellex 50 mg, 2 - 25 mg capsules daily for 3 months
  Interventions: Drug: Proellex 50 mg
- C Placebo (Placebo Comparator): Placebo, 2 capsules daily for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proellex 25 mg — Proellex 25 mg, 1 - 25 mg capsule and 1 placebo capsule daily for 3 months
  Arms: A 25 mg
Drug: Proellex 50 mg — Proellex 50 mg, 2 - 25 mg capsules daily for 3 months
  Arms: B 50 mg
Drug: Placebo — Placebo, 2 capsules daily for 3 months
  Arms: C Placebo

SUMMARY:
Eligible female subjects will be randomly assigned to one of the three treatment groups. Subjects will receive 325 mg (65 mg elemental iron) iron supplements to be taken twice daily during study drug treatment. The study duration is approximately six months, which is comprised of a 4 - 6 week screening period, a three-month drug treatment period, and a one-month follow-up period.

DETAILED DESCRIPTION:
Eligible female subjects will be randomly assigned to one of the three treatment groups. Subjects will receive 325 mg (65 mg elemental iron) iron supplements to be taken twice daily during study drug treatment. The study duration is approximately six months, which is comprised of a 4 - 6 week screening period, a three-month drug treatment period, and a one-month follow-up period.

Study was terminated by clinical hold.

ELIGIBILITY:
Inclusion Criteria:

* Female, between the ages of 18 and 48 years with Body Mass Index (BMI) between 18 and 39, inclusive;
* Anemic, defined as hemoglobin levels less than or equal to 10.5 g/dL and uterine fibroid-associated symptoms indicated by a history of excessive menstrual bleeding;
* Surgical interventions for uterine fibroids (e.g. hysterectomy or myomectomy) planned or anticipated after the study;
* Willing to comply with all study procedures, including the endometrial biopsies and blood draws for all visits, including Follow-up Visits

Exclusion Criteria:

* Post-menopausal women or women likely to become post-menopausal during the study, defined as one or more of the following:

  * Six months or more (immediately prior to Screening Visit) without a menstrual period, or
  * Prior hysterectomy, or
  * Prior bilateral oophorectomy (unilateral oophorectomy is not exclusionary if regular menstruation is occurring);
* Females who have undergone a uterine arterial embolization, or endometrial ablation therapy (previous myomectomy is acceptable) for any cause;
* Documented endometriosis or active pelvic inflammatory disease (PID);
* Having a diagnosis, or suspected diagnosis, of carcinoma of the breast or reproductive organs;
* Known active infection with HIV, Hepatitis A, B or C, Gonorrhea, or Chlamydia;
* Use of prohibited concomitant medications:

  1. Depo-Provera use must cease ten months prior to first dose of study drug, or
  2. GnRH agonists use (e.g. Lupron Depot) must cease six months prior to first dose of study drug, or
  3. Oral contraceptive or other hormonal treatments use must cease for 30 days prior to the start of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre vanAs, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (30):
- United States (30):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Impact Clinical Trials, Los Angeles, California
  - National Institute of Clinical Research, Los Angeles, California
  - Downtown Women's Health Care, Denver, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - OB-GYN Associates of Mid-Florida, P.A., Leesburg, Florida
  - Segal Institute for Clinical Research, Miami, Florida
  - Insignia Clinical Research (Tampa Bay Women's Center), Tampa, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Phoenix Women's Center (eCast), College Park, Georgia
  - Clinical Trials Select (ecast), Decatur, Georgia
  - Dekalb Gynecology Associates/Legacy Obstetrics & Gynecology (eCast), Decatur, Georgia
  - Medical Network for Education and Research, Decatur, Georgia
  - Smith & Hackney, Morrow, Georgia
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Clinical Trials Select (ecast), Silver Spring, Maryland
  - Phoenix OB-GYN Associates, LLC, Moorestown, New Jersey
  - Central Brooklyn Medical Group (eCast), Brooklyn, New York
  - Rapid Medical Research, Inc.(Elite), Cleveland, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - SC Clinical Research Center, Columbia, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Advanced Research Associates, Corpus Christi, Texas
  - Advances in Health Inc., Houston, Texas
  - The Women's Hospital of Texas, Clinical Research Center, Houston, Texas
  - Centex Research, Houston, Texas
  - Institute for Women's Health, San Antonio, Texas
  - Seven Oaks Women's Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- All Groups: Proellex 25 mg, 50 mg or placebo
Period: Overall Study
Arm/Group | All Groups
Started | 56
Completed | 0
Not Completed | 56
Not completed — Study prematurely terminated | 56

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated for safety reasons
Groups:
- 25 mg: Proellex 25 mg, 1 - 25 mg capsule and 1 placebo capsule daily for 3 months
- 50 mg: Proellex 50 mg, 1 - 50 mg capsule and 1 placebo capsule daily for 3 months
- Placebo: Placebo, 2 placebo capsules daily for 3 months
- Total: Total of all reporting groups
Arm/Group | 25 mg | 50 mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin vs Placebo
Description: Comparison between 50 mg Proellex and placebo of change in hemoglobin at month 3
Time Frame: 3 months
Population: Study prematurely terminated for safety reasons
Arm/Group | 25 mg | 50 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Until 1 month after end of treatment, 4 months total.
Description: No adverse event data is available.
Arm/Group | A 25 mg | B 50 mg | C Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights